CLINICAL TRIAL: NCT06776120
Title: The Performance of Fecal Immunochemical Test (FIT) in Diagnosing Colorectal Cancer Among Vietnamese Patients with Lower Gastrointestinal Symptoms
Brief Title: Fecal Immunochemical Test in Diagnosing Colorectal Cancer Among Vietnamese Patients with Lower Gastrointestinal Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luu Ngoc Mai (Other)
Collaborators: Department of Science and Technology, Ho Chi Minh City, Viet Nam (Unknown)
Responsible Party: Sponsor-Investigator, Luu Ngoc Mai, University of Medicine and Pharmacy at Ho Chi Minh City, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3412/DHYD-HDDD
Record Dates: First submitted 2024-12-31; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vietnamese individuals with lower gastrointestinal symptoms (Other): Vietnamese patients aged 40 - 75 years with lower GI symptoms (patients who have experienced at least one month of any lower GI symptoms: lower abdominal pain, constipation, diarrhea, changes in stool caliber, and abdominal bloating) who are examined at the Outpatient Department of the University Medical Center in Ho Chi Minh City or at the Outpatient Department of Nhan Dan Gia Dinh Hospital, Ho Chi Minh City, Vietnam, and are indicated to undergo a first-time screening colonoscopy, will be invited to participate in the study.
  Eligible participants will be instructed to collect their two stool samples within seven days before undergoing bowel preparation. These stool samples will be then submitted for a quantitative FIT (OC-SENSOR, EIKEN CHEMICAL, Japan). Colonoscopic observations and histopathological findings will be employed as the definitive reference standards for diagnosis.
  Interventions: Diagnostic Test: Fecal chemical test (FIT)

INTERVENTIONS:
Diagnostic Test: Fecal chemical test (FIT) — Eligible participants will be instructed to collect their two stool samples within seven days prior to undergoing bowel preparation. These stool samples will be then submitted for a quantitative FIT (OC-SENSOR, EIKEN CHEMICAL, Japan). Colonoscopic observations and histopathological findings will be employed as the definitive reference standards for diagnosis.

SUMMARY:
The goal of this clinical trial is to evaluate the diagnostic value of fecal immunochemical tests (FIT) in identifying colorectal cancer (CRC) among Vietnamese individuals presenting with lower gastrointestinal symptoms.

The main questions it aims to answer are:

1. Does a quantitative FIT with a positive threshold of 10 µg/g effectively diagnose CRC in symptomatic Vietnamese individuals using one and two stool samples?
2. Does combining FIT results with the Asia-Pacific Colorectal Screening (APCS) score improve the diagnostic accuracy for CRC in symptomatic Vietnamese individuals?
3. What is the optimal quantitative FIT threshold for diagnosing CRC and excluding organic colorectal diseases (advanced colorectal polyps, inflammatory bowel disease, ischemic colitis, ...)?
4. How can a standardized protocol for FIT implementation in Vietnamese symptomatic individuals be developed?
5. What are the knowledge and attitudes related to CRC screening among Vietnamese patients with lower gastrointestinal symptoms?
6. What is the acceptability of FIT as a diagnostic tool among Vietnamese patients with lower gastrointestinal symptoms?

Researchers will evaluate the diagnostic performance of FIT with and without the APCS score to determine the optimal approach for identifying patients requiring colonoscopy.

Participants will:

* Provide two stool samples for quantitative FIT.
* Complete a questionnaire assessing clinical and demographic factors, as well as their knowledge, attitudes toward CRC screening, and acceptability of FIT.
* Undergo diagnostic colonoscopy to confirm the presence or absence of colorectal diseases.

This study aims to enhance CRC diagnostic strategies and establish FIT as a widely acceptable and non-invasive diagnostic tool in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria: In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Aged 40 - 75 years.
* Informed consent available.
* Patients with lower GI symptoms (patients who experience at least one month of any lower GI symptoms: lower abdominal pain, constipation, diarrhea, changes in stool caliber, and abdominal bloating) who are scheduled for a first-time screening colonoscopy.

Exclusion Criteria: Individuals meeting any of the following exclusion criteria will be excluded from the study:

1. History of chronic inflammatory bowel disease, diverticular disease of the colon, colorectal surgery, polypectomy, colorectal cancer, artificial heart valves, or vascular graft surgery.
2. Previous colorectal diagnostic imaging, including colonoscopy, sigmoidoscopy, computed tomography (CT) colonography, or barium enema.
3. Presence of alarm symptoms, including lower gastrointestinal bleeding (hematochezia or melena), an abdominal mass, or unexplained clinically significant weight loss (loss of more than 5 kg or 5-10% of body weight over the past 6 months).
4. Symptoms or signs of anorectal tumors or anal ulcers.
5. Acute diarrhea lasting ≤14 days.
6. Current use of aspirin, antiplatelet agents, anticoagulants, or nonsteroidal anti-inflammatory drugs (NSAIDs), as these may cause false-positive FIT results.
7. Diagnosis of hereditary colorectal cancer syndromes (e.g., Lynch syndrome or familial adenomatous polyposis).
8. Pregnancy, breastfeeding, or menstruation at the time of the study.
9. Contraindications to colonoscopy.
10. Incomplete colonoscopy due to failure to advance the scope to the cecum or inadequate bowel preparation (Boston Bowel Preparation Scale [BBPS] score <6 or a segment score <2).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1575 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performances of FIT using one and two stool samples in detecting CRC among Vietnamese patients with lower GI symptoms | through study completion, an average of 24 months
  The sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of FIT (with a positive threshold of 10 µg/g) using one and two stool samples to detect colorectal cancer (CRC), as confirmed by colonoscopy and histopathological findings.

SECONDARY OUTCOMES:
The diagnostic performances of FIT using one and two stool samples combined with APCS scores in detecting CRC among Vietnamese patients with lower GI symptoms | through study completion, an average of 24 months
  The sensitivity, specificity, PPV, and NPV of FIT (with a positive threshold of 10 µg/g) using one and two stool samples, combined with the Asia-Pacific Colorectal Screening (APCS) scores, to detect CRC, as confirmed by colonoscopy and histopathological findings.
  The APCS system consists of four variables (age, sex, smoking history, and family history of CRC). The APCS scores range from 0 to 7. Based on the APCS score, participants will be categorized into three groups: average risk (APCS 0 - 1), moderate risk (APCS 2 - 3), and high risk (APCS 4 - 7).
The diagnostic performances of FIT as a 'rule-out' test for significant colorectal diseases (i.e. CRC, advanced colorectal polyps, inflammatory bowel disease, ischemic colitis …) among Vietnamese patients with lower GI symptoms | through study completion, an average of 24 months
  The sensitivity, specificity, NPV, and PPV of FIT (with a positive threshold of 10 µg/g) using one and two stool samples to rule out significant colorectal diseases (e.g., CRC, advanced colorectal polyps, inflammatory bowel disease, ischemic colitis) among Vietnamese patients presenting with lower gastrointestinal symptoms
Optimal FIT threshold for diagnosing CRC in Vietnamese patients with lower GI symptoms | through study completion, an average of 24 months
  The quantitative FIT threshold using one and two stool samples that maximizes the sensitivity and the specificity to detect CRC in Vietnamese patients with lower GI symptoms
Knowledge, attitude related to CRC screening of Vietnamese patients with lower GI symptoms | through study completion, an average of 24 months
  Measured by a questionnaire, and the measuring unit is multiple choice questions.
The acceptability of FIT in Vietnamese patients with lower GI symptoms | through study completion, an average of 24 months
  Measure the level of acceptability of FIT among the study participants using a structured questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No